CLINICAL TRIAL: NCT00037219
Title: A Phase 2, Open-Label, Randomized, Dose-Ranging Study of the Safety and Efficacy of Intravenous Anidulafungin (VER002) in the Treatment of Patients With Invasive Candidiasis
Brief Title: The Safety and Effectiveness of Intravenous Anidulafungin as a Treatment for Patients With Invasive Candidiasis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Vicuron Pharmaceuticals (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VER002-6; A8851018
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Candidiasis
Keywords: Anidulafungin; Candidemia; Invasive Candidiasis
MeSH Terms: conditions — Candidiasis; Candidemia; Candidiasis, Invasive | interventions — Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin, VER002

SUMMARY:
Anidulafungin may be effective for the treatment of invasive Candida infections. The purpose of the study is to find the balance between dose tolerance and effectiveness of several doses for the treatment of United States patients with invasive candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Positive culture plus at least one clinical sign and symptom consistent with invasive candidiasis preferably within 96 hours of the proposed first dose of study drug
* Life expectancy: greater than 72 hours

Exclusion Criteria:

* Pregnant Females
* Treatment with other investigational drug(s) within 4 weeks
* Hypersensitivity to anidulafungin or echinocandin therapy
* Hypersensitivity to Tween 80 (polysorbate 80) or tartaric acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-08; Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Versicor, Inc., King of Prussia, Pennsylvania, United States